CLINICAL TRIAL: NCT03109236
Title: Autologous Endothelial Progenitor Cell Therapy for Reversal of Liver Cirrhosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore General Hospital (Other); Tan Tock Seng Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/00711
Record Dates: First submitted 2017-03-06; First posted 2017-04-12 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: This is a 2 arm randomised study patients with decompensated liver cirrhosis involving 33 patients in each arm. Randomisation will be done by statistician to determine which arm patients will be in (control / treatment).
  Treatment arm:
  Patient will undergo CD133+ cells transplantation at stable compensated state. 5 dose Granulocyte Colony Stimulating Factor (GCSF) will be administered 5 days consecutively before bone marrow harvesting.
  Approximately 250ml of bone marrow will be harvested and subjected to CD133 isolation using clinimacs (Miltenyi Biotec) in a closed system
  Under ultrasound guidance, 50 mls of 50-100 million CD133 cells will be infused directly through transhepatic route into portal venous circulation of the liver over 5 mins.
  Control Arm:
  Patients will receive 5 doses of GCSF
Who Masked: Outcomes Assessor
Masking Description: Blinding will be maintained by investigators performing analysis of the results. Given the invasive procedure of percutaneous transhepatic cannulation, the investigators felt that it will be unethical to perform sham procedure on control arm patients. Both managing doctors and patient will know which arm they are on but where not inevitable, data collection such as quality of life and results interpretation such as histology and laboratory analysis of results will be performed anonymously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patient will undergo CD133+ cells transplantation at stable compensated state.
  5 dose GCSF will be administered 5 days consecutively before bone marrow harvesting.
  Approximately 250ml of bone marrow will be harvested and subjected to CD133 isolation using clinimacs (Miltenyi Biotec) in a closed system.
  Under ultrasound guidance, 50 mls of 50-100 million CD133 cells will be infused directly through transhepatic route into portal venous circulation of the liver over 5 mins.
  Interventions: Drug: GCSF; Procedure: CD133 Cells Transplantation
- Control (Active Comparator): Non-Transplant Arm:
  Patients will receive 5 doses of GCSF
  Interventions: Drug: GCSF

INTERVENTIONS:
Drug: GCSF — 5 doses of GCSF injection will be injected under the skin on the abdomen to mobilize the bone marrow cells.
Procedure: CD133 Cells Transplantation — Endothelial progenitor cells are harvested by CD133+ MACS (magnetic activated cell sorting) sort selection of bone marrow and a minimum of 1x 10^6 and up to 50-100 x 10^6 cells are transplanted to one lobe of the liver via a percutaneous catheter inserted into the portal venous system by percutaneous transhepatic approach for engraftment.
  Other Names: Endothelial Progenitor cells
  Arms: Treatment

SUMMARY:
This proposal translates a hypothesis driven basic research into clinical setting to determine the potential of using autologous CD133+ cells to reverse fibrosis and improve clinical outcome for patients with end stage cirrhosis. This has significant impact on the management of cirrhosis.

DETAILED DESCRIPTION:
This is a 2 arm randomised study patients with decompensated liver cirrhosis involving minimum of 23 and maximum of 33 patients in each arm.

The investigators propose that transplantation of mobilized autologous CD133+ cells harvested from the bone marrow directly into the liver has the ability to replace and regenerate the damaged sinusoidal endothelium as well as normalize macrophage and Natural Killer (NK) cell function. The niche provided by the refenestrated endothelium can polarize the macrophage to antifibrotic phenotype as well as directly inactivate the activated myofibroblast, resulting in reversal of liver fibrosis and improvement in liver function. Transplantation of cells will be via intraportal route delivered by percutaneous cannulation of the portal vein system.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any aetiology but where active disease is controlled
* Childs A/B/C with Child-Pugh score >= 5

And either one of the following:

1. MELD score 10-27
2. Clinically significant portal hypertension as evidenced by gastroesophageal varices or ascites

Exclusion Criteria:

* MELD score >27
* INR>2.5
* HIV
* History of hematological or hepatic malignancy within 5 years from consent
* Other underlying malignancy with <1 year survival
* Presence of systemic diseases that may impact survival within 1 year.
* Listed for liver transplant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of Fibrosis Staging (Ishak) | 3 months
  Improvement of Fibrosis Staging (Ishak) > 1 point
Improvement of liver fibrosis on MRE (magnetic resonance elastography) | 6 months
  Improvement of liver fibrosis on MRE (magnetic resonance elastography) > 2 point
Improvement of MELD (Model of End stage Liver Disease) score or Child Pugh State | 6 months
  Improvement of MELD (Model of End stage Liver Disease) score or Child Pugh State by at least 2 points
Improvement of quantitative fibrosis | 1 year
  Improvement of quantitative fibrosis on histology > 10%

SECONDARY OUTCOMES:
Overall Survival and Improvement | 1 year
  Overall Survival
Overall Improvement in Liver Function Tests | 1 year
  Improvement in Liver Function Tests, especially Total Bilirubin, Albumin and Prothrombin Time
Improvement of Hepatic Venous Pressure | 3 months
  Improvement of Hepatic Venous Pressure
Incidence of clinical decompensation | 1 year
  Frequency of Incidence of clinical decompensation
Overall Improvement of Patient Reported outcome | 6 months
  Improvement of Patient Reported outcome (quality of life Short Form Health Survey SF-36 for liver cirrhosis)
Overall Improvement of MELD score | 1 year
  Rate of deterioration of MELD score (Kaplan Meier analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Yock Young, Principal Investigator — National University Hospital, Singapore; Mark Muthiah, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore